CLINICAL TRIAL: NCT02324283
Title: Comparison of Emergence and Recovery Time, and Evaluation of Oxygenation During One-lung Ventilation With Desflurane and Propofol Anesthesia in Lung Surgery- A Pilot Study
Brief Title: Comparison of Emergence and Oxygenation During One-lung Ventilation With Desflurane and Propofol Anesthesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juntendo University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12-97
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: one-lung ventilation, oxygenation
MeSH Terms: conditions — Lung Neoplasms | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): Desflurane group: this group of patients receives desflurane as the main anesthetic agent in addition to remifentanil infusion at 0.1~0.3 mcg/kg/min during one-lung anesthesia. Bispectral index will be maintained between 45 and 50. Arterial blood gases and pulmonary blood flow by using tansesphageal echocardiogrphy will be measured.
  Interventions: Drug: desflurane
- Propofol (Active Comparator): Propofol group: this group of patients receives propofol as the main anesthetic agent in addition to remifentanil infusion at the rate of 0.1~0.3 mcg./g/min during one-lung anesthesia. Bispectral index will be maintained between 45 and 50. Arterial blood gases and pulmonary blood flow by using tansesphageal echocardiogrphy will be measured.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: desflurane — Desflurane group: this group of patients receives desflurane as the main anesthetic agent during one-lung anesthesia.
  Propofol group: this group of patients receives propofol as the main anesthetic agnet during on-lung anesthesia.
  Other Names: Suprene
  Arms: Desflurane
Drug: propofol — Propofol group:this group of patients receives propofol as the main anesthetic agent during one-lung anesthesia.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
Which is more adequate general anesthetic agent, desflurane or propofol, for emergence and recovery time, and perioperative oxygenation in lung resection surgery?

DETAILED DESCRIPTION:
The investigators plan to investigate the effects of desflurane on oxygenation (prevention of HPV) of OLV compare with propofol which is used in general anesthesia for lung resection.

Transesophageal echocardiography (TEE) wiill be used to measure pulmonary blood flow during surgery visible and successively. To confirm the effect of HPV by measuring the change in pulmonary blood flow. The correlation between the blood oxygen concentration and attenuation of blood flow will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients agree to participate in the study
* Patients undergoing lung cancer surgery requiring one-lung ventilation.
* American Society of Anesthesiologists Physical Status Class 1 or 2

Exclusion Criteria:

* Patients with any of the following will be excluded from lung cancer patients.
* New York Heart Association Classification more than 2
* Respiratory dysfunction Vital Capacity or percent predicted Forced expiratory volume in one second is less than 50 %
* Pulmonary hypertension with mean pulmonary arterial pressure more than 30 mmHg
* Coagulation dysfunction
* The administration of steroids and immunosuppressive agents within 3 months prior to surgery
* Infection with active inflammation
* Pneumonectomy patients
* Cases of epidural anesthesia is contraindicated

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2024-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eiichi Inada, M.D., Principal Investigator — Juntendo University
Locations (1):
- University of Juntendo, Bunkyō City, Tokyko, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Desflurane: Desflurane group: this group of patients receives desflurane as the main anesthetic agent in addition to remifentanil infusion at 0.1~0.3 mcg/kg/min during one-lung anesthesia. Bispectral index will be maintained between 45 and 50. Arterial blood gases and pulmonary blood flow by using tansesphageal echocardiogrphy will be measured.
  desflurane: Desflurane group: this group of patients receives desflurane as the main anesthetic agent during one-lung anesthesia.
  Propofol group: this group of patients receives propofol as the main anesthetic agnet during on-lung anesthesia.
Period: Overall Study
Arm/Group | Desflurane | Propofol
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane | Propofol | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.7) | 63.2 (6.6) | 63.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 21 | 24 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Oxygenation
Description: Arterial blood gases are monitored.Pulmonary blood flow is measured using transesophageal echocardiogram.
Time Frame: prior to surgery to one-hour after extubation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 40 | 40
mmHg
  Preoperative | 87.4 (12.0) | 85.7 (11.3)
  DLV(pre) | 469.9 (79.8) | 483.8 (91.7)
  OLV(15min) | 178.5 (95.0) | 214.7 (114.2)
  OLV(30min) | 137.7 (78.2) | 161.6 (95.4)
  OLV(45min) | 140.7 (86.6) | 171.57 (95.6)
  DLV(post) | 429.9 (98.3) | 427.49 (111.6)
  5min after exT | 131.63 (44.2) | 134.88 (64.0)
  30min after exT | 125.71 (45.3) | 125.65 (32.91)
  60min after exT | 130.49 (45.0) | 137.2 (36.0)

2. Secondary Outcome: Rapidity of Emergence From Anesthesia
Description: Time to extubation and orientation, where the patient is.
Time Frame: one minute after cessation of anethetic agents to one hour after extubation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 40 | 40
seconds | 252.3 (156.3) | 269.5 (142.9)

3. Secondary Outcome: Quality of Consiousness
Description: quality of consciousness will be assessed using Aldrete score
Time Frame: after extubation
Population: number of the patients who cannot achieve full consciousness in Aldlete score 5min after extubation
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 40 | 40
participants | 2 | 0

4. Secondary Outcome: Postoperative Nausea and Vomiting
Description: degree of nausea and frequency of vomiting
Time Frame: on the postoperative day 1
Population: the number of patients who encountered PONV for 24 hours after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 40 | 40
Participants | 15 | 10

ADVERSE EVENTS:
Arm/Group | Desflurane | Propofol
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No